CLINICAL TRIAL: NCT07229729
Title: A Randomized, Open-label, Multicenter Phase II Clinical Study of SHR-A2102 in Combination With Other Anti-tumor Therapies for Perioperative Treatment of Resectable Non-small Cell Lung Cancer
Brief Title: A Study of SHR-A2102 in Combination With Other Anti-tumor Therapies for Resectable Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2102-212
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin; osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A2102 + Adebrelimab + Paclitaxel + Carboplatin Group (Experimental)
  Interventions: Drug: SHR-A2102; Drug: Adebrelimab; Drug: Paclitaxel; Drug: Carboplatin
- SHR-A2102 + Alomnertinib/Osimertinib/Furmonertinib Group (Active Comparator)
  Interventions: Drug: SHR-A2102; Drug: Alomnertinib Mesilate; Drug: Furmonertini Mesilate; Drug: Osimertinib Mesylate

INTERVENTIONS:
Drug: SHR-A2102 — SHR-A2102.
Drug: Adebrelimab — Adebrelimab.
  Arms: SHR-A2102 + Adebrelimab + Paclitaxel + Carboplatin Group
Drug: Paclitaxel — Paclitaxel.
  Arms: SHR-A2102 + Adebrelimab + Paclitaxel + Carboplatin Group
Drug: Carboplatin — Carboplatin.
  Arms: SHR-A2102 + Adebrelimab + Paclitaxel + Carboplatin Group
Drug: Alomnertinib Mesilate — Alomnertinib Mesilate.
  Arms: SHR-A2102 + Alomnertinib/Osimertinib/Furmonertinib Group
Drug: Furmonertini Mesilate — Furmonertini Mesilate.
  Arms: SHR-A2102 + Alomnertinib/Osimertinib/Furmonertinib Group
Drug: Osimertinib Mesylate — Osimertinib Mesylate.
  Arms: SHR-A2102 + Alomnertinib/Osimertinib/Furmonertinib Group

SUMMARY:
The study is a Phase II study to explore the efficacy and safety of SHR-A2102 in combination with other anti-tumor therapies as perioperative treatment in patients with resectable non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this clinical study, understand the research procedures and be able to sign the informed consent form in writing;
2. Participants must be aged between 18 and 70 years old (inclusive) when signing the informed consent form, and both men and women are eligible;
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
4. Adequate organ function;
5. Women of childbearing age must undergo serum pregnancy tests, and the results must be negative. Female subjects of childbearing age and male subjects who are partners of women of childbearing age must agree to use highly effective contraceptive methods.

Exclusion Criteria:

1. With active, known or suspected autoimmune disease of autoimmune disease;
2. Malignancies other than NSCLC within 5 years prior to randomization;
3. Has or suspected has a history of pneumonitis / interstitial lung disease or any serve lung diseases which will influence the examination of lung function;
4. Significant history of cardiovascular and cerebrovascular disease; Significant haemorrhagic disease;
5. Has an arteriovenous thrombotic events;
6. Has a known history of human immunodeficiency virus (HIV) infection;
7. Has a known active Hepatitis B or Hepatitis C;
8. Allergic to the intervention regimens.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Pathology complete response (pCR) | Up to approximately 20 weeks.
18-month event free rate | Up to approximately 18 months.
2-years disease free rate | Up to approximately 2 years.

SECONDARY OUTCOMES:
Event free survival (EFS) | Up to approximately 5 years.
Overall survival (OS) | Up to approximately 5 years.
Objective response rate (ORR) | Up to approximately 20 weeks.
Disease-Free Survival (DFS) | Up to approximately 5 years.
Adverse events (AEs) | Up to approximately 5 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided